CLINICAL TRIAL: NCT01718678
Title: Study of Melatonin in Treatment of Fatigue in Multiple Sclerosis
Brief Title: Effect of Melatonin on Multiple Sclerosis Related Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Shemshaki, research assistant, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-12111
Record Dates: First submitted 2012-10-28; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Fatigue
Keywords: Multiple sclerosis; Melatonin; Fatigue; Quality of life
MeSH Terms: conditions — Fatigue; Multiple Sclerosis | interventions — Melatonin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Active Comparator): Melatonin, Tablet, 3 mg, once, one month
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo, tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — it is kind of drug
  Arms: Melatonin
Drug: Placebo — It is Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of Melatonin in treatment of fatigue and Quality of Life of MS patients.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is one of the most common non-traumatic causes of disability in the world. It is a chronic inflammatory and demyelinating disorder of the Central Nervous System (CNS) which affects individuals in the productive ages and causes a large burden for years to come. Fatigue is a common complaint and one of the least understood symptoms of MS

ELIGIBILITY:
Inclusion Criteria:

1. definite diagnosis of relapsing-remitting MS (RRMS) by the MacDonald criteria
2. a baseline of Expanded Disability Status Score (EDSS)of less than 5.0
3. aged between 18 and 55 years of either sex
4. treated with one type of interferon beta-1a (IFNB-1a);
5. signed an informed consent

Exclusion Criteria:

1. clinical relapsing of MS during past 30 days;
2. use of melatonin and warfarin within 30 days prior to participation;
3. concomitant use of beta-blockers, anti-diabetic agents, antiplatelet agents, NSAIDS, aspirin ;
4. working more than one nighttime shift per month;
5. Pregnancy or lactation;
6. history of a chronic hematological, cardiac, hepatic, renal or thyroid disorders ;
7. failure to adhere to the study protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Fatigue | at one month after treatment
  Modified Fatigue Impact Scale (MFIS)is a21-item (score range of each item: 0-4) questionnaire with the total score computed from 0 (no impact of fatigue) to 84 (maximum impact of fatigue) in three subscales containing: physical (9 items), cognitive (10 items) and psychosocial (2 items) aspects.

SECONDARY OUTCOMES:
Quality Of Life | at one month after treatment
  Quality Of Life Questionnaire (MSQOL-54) consisted of 54 questions (items), each one, assigned to a score ranging from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran